CLINICAL TRIAL: NCT02664571
Title: Evaluation of Florbetaben as an Amyloid Plaque Marker in Elderly Patients With Focal or Disseminated Superficial Hemosiderosis
Brief Title: Florbetaben as an Amyloid Plaque Marker in Elderly Patients With Focal or Disseminated Superficial Hemosiderosis
Acronym: FBB ACC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: experimental drug prohibited by the ANSM (French competent authority)
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LOCAL/2015/DM-01; 2015-004583-11 (EudraCT Number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Amyloid Cerebral Angiopathy; Alzheimer Disease
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Alzheimer Disease | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ACA with isolated hemosiderosis (Other): This group is composed of patients with amyloid cerebral angiopathy (ACA) with isolated hemosiderosis.
  Intervention: Pet scan with FBB
  Intervention: MRI scan
  Intervention: APO E genotyping
  Interventions: Device: Pet scan with FBB; Device: MRI scan; Biological: APO E genotyping
- ACA with lobar hematoma(s) (Other): This group is composed of patients with amyloid cerebral angiopathy (ACA) with lobar hematoma(s).
  Intervention: Pet scan with FBB
  Intervention: MRI scan
  Intervention: APO E genotyping
  Interventions: Device: Pet scan with FBB; Device: MRI scan; Biological: APO E genotyping
- Alzheimer's without ACA (Other): This group is composed of Alzheimer's type dementia without MRI signs in favor of amyloid cerebral angiopathy (ACA).
  Intervention: Pet scan with FBB
  Intervention: MRI scan
  Intervention: APO E genotyping
  Interventions: Device: Pet scan with FBB; Device: MRI scan; Biological: APO E genotyping
- Healthy volunteers (Other): This group is composed of healthy volunteers.
  Intervention: Pet scan with FBB
  Intervention: MRI scan
  Intervention: APO E genotyping
  Interventions: Device: Pet scan with FBB; Device: MRI scan; Biological: APO E genotyping

INTERVENTIONS:
Device: Pet scan with FBB — Patients will have a pet scan with Florbetaben (NEURACEQ : FBB). All other care corresponds to routine care.
  Florbetaben is used during pet scans to visualize beta amyloid plaques and cannot be a separate intervention in and of itself.
Device: MRI scan — Subjects will have an MRI scan at inclusion.
Biological: APO E genotyping — Subjects will have APO (apolipoprotein) E genotyping if not already known.

SUMMARY:
The main objective of this study is to compare the distribution of Florbetaben (NEURACEQ: FBB) in the brain in amyloid cerebral angiopathy (ACA) manifested by isolated hemosiderosis in non-demented patients with that observed in healthy subjects, patients with ACA and with lobar hematoma(s) and patients with Alzheimer's dementia without MRI signs in favor of ACA.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare among groups:

A. The associated micro-bleeds. B. Associated leukoencephalopathy. C. Contrast observed in lobar Virchow-Robin perivascular spaces. D. Apolipoprotein E genotypes.

ELIGIBILITY:
Inclusion Criteria for patients with amyloid cerebral angiopathy with isolated hemosiderosis:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has a single or multiple focal spontaneous hemosiderosis objectified by an MRI
* The patient is does not have dementia (Mini Mental State score> 27)

Inclusion Criteria for patients with amyloid cerebral angiopathy with with lobar hematoma(s):

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has one or more spontaneous lobar hematomas with or without hemosiderosis objectified by an MRI
* The patient is does not have dementia (Mini Mental State score> 27)

Inclusion Criteria for patients with Alzheimer's type dementia without MRI signs in favor of amyloid cerebral angiopathy:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has Alzheimer's dementia (Mini Mental State score <24) without hemosiderosis or previous lobar hematoma or history of other brain lesion seen on MRI

Inclusion Criteria for health volunteers:

* The subject must have given his/her informed and signed consent
* The subject must be insured or beneficiary of a health insurance plan
* Healthy volunteers without cerebral neurological history and with normal MRI
* The subject is does not have dementia (Mini Mental State score> 27)

Exclusion Criteria for patients with amyloid cerebral angiopathy with isolated hemosiderosis:

* The patient is participating in another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The subject (next of kin or legal representative) refuses to sign the consent
* It is not possible to give the subject or his/her representative informed information
* The patient has an contra-indication for performing an MRI
* The patient is in the acute phase (the tracer does not bind in cases of large hematoma)

Exclusion Criteria for patients with amyloid cerebral angiopathy with with lobar hematoma(s):

* The patient is participating in another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The subject (next of kin or legal representative) refuses to sign the consent
* It is not possible to give the subject or his/her representative informed information
* The patient has an contra-indication for performing an MRI
* The patient is in the acute phase (the tracer does not bind in cases of large hematoma)

Exclusion Criteria fpr patients with Alzheimer's type dementia without MRI signs in favor of amyloid cerebral angiopathy:

* The patient is participating in another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The subject (next of kin or legal representative) refuses to sign the consent
* It is not possible to give the subject or his/her representative informed information
* The patient has an contra-indication for performing an MRI
* The patient is in the acute phase (the tracer does not bind in cases of large hematoma)
* Haemosiderosis or history of lobar hematoma or other visible cerebral history on MRI

Exclusion Criteria for healthy volunteers:

* The subject is participating in another interventional study
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection
* The subject (next of kin or legal representative) refuses to sign the consent
* It is not possible to give the subject or his/her representative informed information
* The subject has an contra-indication for performing an MRI
* Abnormal MRI

The groups will be matched according to sex and age (by increments of 5 years) to the extent possible. Because amyloid cerebral angiopathy is a very rare condition, matching the two factors may be difficult to achieve. We therefore anticipate where appropriate to focus matching on age.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
PET scan with Florbetaben: Standardized Uptake Value Ratio | Day 0

SECONDARY OUTCOMES:
On the reference MRI: the number of lobar hemorrhages | Day 0
On the reference MRI: the locations of lobar hemorrhages | Day 0
  Location is defined as choices from among the following: frontal-right; frontal-left; parietal-right; parietal-left; occipital-right; occipital-left; temporal-right; temporal-left.
On the reference MRI: The presence/absence classification for superficial siderosis | Day 0
  The classification corresponds to one of the following: absence; focal (involving < 4 sulci); disseminated (involving 4 or more sulci).
On the reference MRI: the locations of superficial siderosis | Day 0
  Location is defined as choices from among the following: frontal-right; frontal-left; parietal-right; parietal-left; occipital-right; occipital-left; temporal-right; temporal-left.
On the reference MRI: the absolute quantitative count of microbleeds | Day 0
On the reference MRI: microbleed count category | Day 0
  The microbleed count category corresponds to one of the following: 0, 1, 2-4, >4.
On the reference MRI: The predominant location of microbleeds | Day 0
On the reference MRI: a measure of leukoencephalopathy using the ARWMC scale | Day 0
  The age-related white matter changes (ARWMC) rating scale rating only the supratentorial white matter for each frontal, parieto-occipital, and temporal localisation: 0 for no lesions, 1 for focal lesions, 2 for beginning confluence of lesions, and 3 for diffuse involvement of the entire region
Apolipoprotein E genotype | Day 0
  Everyone has two copies of the gene so the resulting combination determines your APOE "genotype" as one of the following: E2/E2, E2/E3, E2/E4, E3/E3, E3/E4, or E4/E4.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Renard, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CH de Perpignan - Hôpital Saint Jean, Perpignan